CLINICAL TRIAL: NCT00815178
Title: Effects of Inspiratory Muscle Training on Type 2 Diabetes Mellitus Patients With Inspiratory Muscle Weakness: A Randomized, Controlled Clinical Trial
Brief Title: Effects of Inspiratory Muscle Training on Type 2 Diabetes Mellitus Patients With Inspiratory Muscle Weakness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Inspiratory training diabetes
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Last update posted 2008-12-29 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes Complications; Inspiratory Muscle Weakness
Keywords: inspiratory muscle weakness; autonomic modulation; diabetes mellitus; heart rate variability; functional capacity
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory muscle training (Experimental)
  Interventions: Behavioral: Inspiratory muscle training
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Inpiratory muscle training placebo

INTERVENTIONS:
Behavioral: Inspiratory muscle training — For Inspiratory muscle training (IMT)patients carried out the IMT on a daily basis for eight weeks, with duration of 30 minutes and intensity corresponding to 30% of resting PImax, with a linear pressure resistance device (Threshold®). Weekly maximum inspiratory pressure (PImax) evaluations and workload adjustments were performed. Inspiratory load was adjusted on a weekly basis to maintain 30% of the subject's PImax. Training sessions were carried out at home for both groups and supervised once a week at the hospital.
  Arms: Inspiratory muscle training
Behavioral: Inpiratory muscle training placebo — Inspiratory muscle training was carried out on the same basis as in the intervention group but with no inspiratory load.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if inspiratory muscle training improves inspiratory muscle strength of type 2 diabetes mellitus patients with inspiratory muscle weakness.

DETAILED DESCRIPTION:
In congestive heart failure patients, inspiratory muscle weakness can be reversed by developing diaphragmatic hypertrophy through inspiratory muscle training, improving functional capacity and quality of life. In type 2 diabetes mellitus patients the frequency of inspiratory muscle weakness is unknown, as well as the response to inspiratory muscle training. For this reason, the present study evaluated the inspiratory muscle strength in type 2 diabetes mellitus patients and the effect of inspiratory muscle training on inspiratory muscle strength, pulmonary function, functional capacity and autonomic modulation assessed through heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* diabetes melittus
* sedentary
* inspiratory muscle weakness with PImax < 70% of the predicted

Exclusion Criteria:

* mass index > 33 kg/m2
* exercise-induced asthma history
* infectious disease
* osteoarticular disease
* regular alcohol or tobacco consumption in the past 6 months
* cardiac disease
* pulmonary disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory pressure | 8 weeks

SECONDARY OUTCOMES:
Peak exercise oxigen consumption | 8 weeks
pulmonary function | 8 weeks
autonomic modulation assessed by heart rate variability | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Chiappa GR, Roseguini BT, Vieira PJ, Alves CN, Tavares A, Winkelmann ER, Ferlin EL, Stein R, Ribeiro JP. Inspiratory muscle training improves blood flow to resting and exercising limbs in patients with chronic heart failure. J Am Coll Cardiol. 2008 Apr 29;51(17):1663-71. doi: 10.1016/j.jacc.2007.12.045. PMID 18436118
- [Derived] Correa AP, Ribeiro JP, Balzan FM, Mundstock L, Ferlin EL, Moraes RS. Inspiratory muscle training in type 2 diabetes with inspiratory muscle weakness. Med Sci Sports Exerc. 2011 Jul;43(7):1135-41. doi: 10.1249/MSS.0b013e31820a7c12. PMID 21200342